CLINICAL TRIAL: NCT01137539
Title: TVT-SECUR as an Office-based Procedure - A Pilot Study
Brief Title: TVT-SECUR as an Office-based Procedure
Acronym: TVTSOffice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan Institution of Women's Health PC (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Salil Khandwala MD, President, Michigan Institution of Women's Health PC, Michigan Institution of Women's Health PC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIWH08-001
Record Dates: First submitted 2010-05-24; First posted 2010-06-04 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Urinary Incontinence; Stress Urinary Incontinence
Keywords: urinary incontinence; stress urinary incontinence; mid-urethral slings; Tension-free vaginal taping; TVT
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gynecare TVT-SECUR system (Experimental): All patients enrolled into the study will receive the TVT-SECUR system to treat stress urinary incontinence
  Interventions: Device: Gynecare TVT-SECUR system

INTERVENTIONS:
Device: Gynecare TVT-SECUR system — All patients in the study will receive the Gynecare TVT-SECUR to treat stress urinary incontinence
  Other Names: TVT-S; Mid-urethral sling

SUMMARY:
This is a pilot study to assess the feasibility and success of performing the TVT-Secur in the office setting. Endpoints would be success, complications, and patient and physician acceptance of the procedure. Success would be assessed by validated questionnaires.

This is a prospective single arm study of 50 patients who will have the TVT-Secur procedure done in the office under local anesthesia. They will be followed for a period of 3 years.

DETAILED DESCRIPTION:
The study will include 50 patients who would meet the inclusion/exclusion criteria and who sign the informed consent. Subjects are diagnosed with Stress urinary incontinence resulting from urethral hypermobility with no prior urinary incontinence surgery. Subjects are women who no longer intend to bear children and who do not require any other concomitant surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence with hypermobility of the UV junction
* ASA I or II
* Age 21-89

Exclusion Criteria:

* Prior anti-incontinence surgery
* Not completed childbearing
* ASA III or higher
* Need concomitant surgery
* Poor compliance for office based approach

Ages: 21 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salil S Khandwala, MD, Principal Investigator — Michigan Institute of Women's Health PC
Locations (1):
- Advanced Urogynecology of Michigan PC, Dearborn, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: October 2008-May 2009 at medical practice
Period: Overall Study
Arm/Group | Gynecare TVT-SECUR System
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gynecare TVT-SECUR System
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 1
Age, Continuous [Median (Standard Deviation); unit: years] | 46.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47
  Hispanic or Latino | 3
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Based on Patient Report on Validated Questionnaire
Description: Negative response to question #3 on the Urogenital Distress Inventory-6 (UDI-6) questionnaire. Question #3 states, "Do you currently experience urine leakage related to physical activity, coughing or sneezing." If a subject answers "No", this is considered success. If a subject answers "Yes", this is considered failure of treatment.
Time Frame: 24 months
Population: 46 subjects were analyzed at the 24 month period out of the total 50 subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecare TVT-SECUR System
Number analyzed (Participants) | 46
Participants | 42

2. Secondary Outcome: Patient Satisfaction
Description: Positive response to a satisfaction question
Time Frame: 12 months
Population: 49 subjects were analyzed at the 12 month period out of the total 50 subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecare TVT-SECUR System
Number analyzed (Participants) | 49
Participants | 47

ADVERSE EVENTS:
Time Frame: Adverse event data collected for 36 months following subject TVT-Secur procedure date.
Arm/Group | Gynecare TVT-SECUR System
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 1/50
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gynecare TVT-SECUR System (N=50)
Mesh Exposure (Product Issues) | 1 — 1 cm x 1 cm mesh exposure noted during follow-up examination. This was managed expectantly by the principal investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes